CLINICAL TRIAL: NCT01611935
Title: AVERT Shock: Arginine Vasopressin During the Early Resuscitation of Traumatic Shock
Acronym: AVERTShock
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Trauma Research Institute (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 811293
Record Dates: First submitted 2012-06-01; First posted 2012-06-05 (Estimated); Results first posted 2019-05-21 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-04

CONDITIONS: Traumatic Shock
Keywords: trauma; shock; vasopressin; blood transfusion
MeSH Terms: conditions — Shock, Traumatic; Wounds and Injuries; Shock; Diabetes Insipidus | interventions — Vasopressins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vasopressin (Active Comparator): Vasopressin will be given as an initial bolus (4 Units) followed by an infusion titrated between 0 units/min to 0.04 units per min to maintain a mean arterial blood pressure greater than or equal to 65 mmHg
  Interventions: Drug: Vasopressin
- Normal Saline (Placebo Comparator): An initial bolus of normal saline will be given (10 cc) and an infusion of 0.1 ml per minute will be started and titrated down in as the mean arterial blood pressure reaches 65 mmHg or more.
  Interventions: Drug: Vasopressin

INTERVENTIONS:
Drug: Vasopressin — After receiving greater than 6 units of blood product within the first 12 hours of admission, trauma patients will be randomized to either normal saline or vasopressin. Subjects will receive an initial 4 unit bolus followed by an infusion of 0 to 0.04 units titrated to maintain a mean arterial blood pressure of equal to or greater than 65 mmHg for a total of 48 hours.

SUMMARY:
Trauma patients, who are transfused with multiple blood products to treat shock due to blood loss, frequently develop inappropriately low vasopressin levels. Vasopressin is a hormone necessary to maintain an adequate blood pressure and low levels have been associated with the need for increased transfusions, vasopressors and additional morbidity. Vasopressin is routinely used in the ICU to treat septic shock and other disease processes resulting in decreased vasopressin levels and low blood pressure. This study will investigate the potential benefit of early vasopressin supplementation during the resuscitation of trauma patients and the applicability of using copeptin as a vasopressin biomarker. Trauma patients who receive 6 or more units of blood product within 12 hours of arrival will be randomized to receive a vasopressin bolus plus infusion or a similar volume of a placebo (normal saline) for 48 hours. Serial blood samples will be taken for 5 days post-injury. Clinical and demographic data will be recorded prospectively.

DETAILED DESCRIPTION:
Trauma remains the leading cause of death for those under the age of 40 in the United States, with a large percentage of patients dying from blood loss within the initial post-injury hours. Although resuscitation with intravenous fluids and blood products has remained the gold standard over the last twenty years, vigorous volume resuscitation may not be curative and has been associated with the development of serious complications including coagulopathy, acute lung injury, and abdominal compartment syndrome. Massive resuscitation also profoundly alters the neuroendocrine milieu needed to maintain vasomotor tone and these severely injured patients may progress to a state of recalcitrant hypotension, multi-organ failure, and ultimately death. The inclusion of vasoactive hormones during resuscitation could potentially prevent the profound hypotension seen in late stage shock, limit the need for aggressive volume and blood product resuscitation, and decrease the incidence of resuscitation-associated complications. As such, there exists an urgent need to evaluate novel resuscitation strategies that target neuroendocrine deficiencies in hemorrhagic shock. The hormone arginine vasopressin (AVP), in particular, may prove a useful adjunct during resuscitation. Secreted by the posterior pituitary, vasopressin is essential for maintaining vasomotor tone during hemorrhagic shock and low levels are associated with the development of catecholamine-resistant hypotension and profound venodilation. Trauma patients who require more than 5 units of blood products during their initial resuscitation are at risk for developing a vasopressin insufficiency, the need for vasopressor support, and often require longer ICU stays. Vasopressin has enjoyed widespread off-label use as a vasopressor in cardiac arrest, septic shock, and post-cardiopulmonary vasodilatory shock. The central hypothesis is that trauma patients who present in hemorrhagic shock are at risk for vasopressin deficiency and would benefit from early vasopressin supplementation. This study will investigate if early use of vasopressin during the resuscitation of traumatic shock results in fewer blood transfusions, a decreased need for crystalloid resuscitation, and a lower incidence of resuscitation related complications.

ELIGIBILITY:
Inclusion Criteria:

* Trauma patients between the ages of 18 and 65 who require 6 or more units of blood product during their initial 12 hours of resuscitation will be considered for enrollment.

Exclusion Criteria:

* Patients with a traumatic brain injury requiring neurosurgical operative intervention or who have neurologic trauma deemed non-survivable will also be excluded.
* Patients with an active coronary syndrome, history of myocardial infarction or coronary artery disease will be excluded.
* Patients with known renal dysfunction requiring dialysis will be excluded.
* Patients who are pregnant will be excluded.
* Patients less than 18 years old will be excluded.
* Patients who have opted out by bracelet identification or by listing themselves on the "Non-Participant" roster.
* Patients under the jurisdiction of the department of corrections and considered prisoners prior to the initiation of the research intervention will be excluded

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2016-09-06 (Actual); Study Completion 2016-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carrie A Sims, MD, MS, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital at the Unversity of Pennyslvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sims CA, Holena D, Kim P, Pascual J, Smith B, Martin N, Seamon M, Shiroff A, Raza S, Kaplan L, Grill E, Zimmerman N, Mason C, Abella B, Reilly P. Effect of Low-Dose Supplementation of Arginine Vasopressin on Need for Blood Product Transfusions in Patients With Trauma and Hemorrhagic Shock: A Randomized Clinical Trial. JAMA Surg. 2019 Nov 1;154(11):994-1003. doi: 10.1001/jamasurg.2019.2884. PMID 31461138

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vasopressin | Normal Saline
Started | 50 | 51
Completed | 49 | 51
Not Completed | 1 | 0
Not completed — Family Declined Participation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vasopressin | Normal Saline | Total
Number analyzed (Participants) | 49 | 51 | 100
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 26 [21 to 31] | 27 [24 to 36] | 26 [23 to 34]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 46 | 47 | 93
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 42 | 40 | 82
  White | 7 | 8 | 15
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 49 | 51 | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Blood Products Transfused
Description: Cumulative number of units of blood products, including packed red blood cells, plasma and platelets measured in liters
Time Frame: 48 hours following the initiation of therapy
Measure: Median (Inter-Quartile Range); unit: Litre
Arm/Group | Vasopressin | Normal Saline
Number analyzed (Participants) | 49 | 51
Litre | 1.7 [0.7 to 3.1] | 3.0 [1.4 to 5.2]

2. Secondary Outcome: Need for Vasopressor Requirement Vasopressor Requirement
Description: total dose of vasopressors (epinephrine, norepinephrine, neosynephrine, etc) received by patient within 48 hours converted to norepinephrine equivalents (g) range in our study was from 0 gm to a max of 53 gm
Time Frame: 48 hours following the initiation of therapy
Measure: Median (Inter-Quartile Range); unit: Norepinephrine equivalents (g)
Arm/Group | Vasopressin | Normal Saline
Number analyzed (Participants) | 49 | 51
Norepinephrine equivalents (g) | 0.6 [0 to 14] | 1.5 [0.2 to 14]

3. Secondary Outcome: Total Number of Complications
Description: Variables will include intra-abdominal hypertension, open abdomen free days, ventilator-free days, ICU-free days, development of ARDS, development of renal failure, development of multiple organ failure, volume of crystalloid requirement within 48 hours post injury, and mortality.
Time Frame: 30 days post injury
Population: patients who did not survive the 48 hours were not included in the analysis
Measure: Number; unit: Complications
Arm/Group | Vasopressin | Normal Saline
Number analyzed (Participants) | 44 | 47
Complications | 69 | 98

ADVERSE EVENTS:
Time Frame: 30 days post enrollment
Arm/Group | Vasopressin | Normal Saline
All-Cause Mortality (participants affected / at risk) | 5/49 | 4/51
Serious Adverse Events (participants affected / at risk) | 30/49 | 36/47
Other Adverse Events (participants affected / at risk) | 22/44 | 28/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Vasopressin (N=49) | Normal Saline (N=47)
Acute Renal Failure (Renal and urinary disorders) | 2/44 (2) | 8 (8)
ARDS (Respiratory, thoracic and mediastinal disorders) | 29/44 (29) | 36 (36)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vasopressin (N=44) | Normal Saline (N=47)
Deep Venous Thrombosis (Blood and lymphatic system disorders) | 5 (5) | 16 (16)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 7 (7) | 7 (7)
Wound Infection (Infections and infestations) | 4 (4) | 5 (5)
Sepsis (Infections and infestations) | 2 (2) | 6 (6)
Extremity Compartment Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Hyponatremia (Renal and urinary disorders) | 5 (5) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No